CLINICAL TRIAL: NCT00755482
Title: Randomised, Placebo Controlled Trial to Examine the Effect of Aquamin F on NSAID Dose Reduction in Subjects With Osteoarthritis of the Knee.
Brief Title: Effects of Aquamin F on NSAID Dose Reduction in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Marigot Ltd. (Industry)
Responsible Party: Marigot Ltd
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MARC005-080
Record Dates: First submitted 2008-09-18; First posted 2008-09-19 (Estimated); Last update posted 2008-09-19 (Estimated); Status verified 2008-09

CONDITIONS: Osteoarthritis of the Knee
Keywords: Osteoarthritis; Clinical trial; Aquamin F; NSAID
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Subjects were given Aquamin F
  Interventions: Drug: Aquamin F
- 2 (Placebo Comparator): Subjects were given a maltodextran placebo
  Interventions: Drug: Placebo (maltodextran)

INTERVENTIONS:
Drug: Aquamin F
  Arms: 1
Drug: Placebo (maltodextran)
  Arms: 2

SUMMARY:
The objective of this trial is to evaluate the effect of Aquamin F versus placebo on NSAID (non-steroidal anti-inflammatory drug) dose reduction in subjects with osteoarthritis of the knee.

Hypothesis 1: After 12 weeks of treatment, subjects taking Aquamin F will use significantly less NSAID medications for symptoms of osteoarthritis versus placebo alone.

Hypothesis 2: No significant differences will be seen for adverse events between the subjects taking Aquamin F or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 35 to 75, male or female
* Subjects diagnosed with symptomatic moderate to severe osteoarthritis of the knee according to the modified criteria of the American College of Rheumatology 17,18
* Subjects who present with osteoarthritis of the knee as judged by symptoms and disabilities detectable through published, validated questionnaires or previous diagnosis by a physician
* subjects who are symptomatic with daily or near daily pain and stiffness from osteoarthritis
* subjects who are taking non-steroidal anti-inflammatory drugs (NSAIDs) prior to study enrollment
* subjects who are willing to stop NSAIDS and use acetaminophen for pain management during the trial
* subjects with screening WOMAC osteoarthritis index total score (transformed score) of not more than 75
* subjects with ability to comprehend and complete the questionnaires and forms
* subjects whose schedules permit clinical evaluations every four weeks
* subjects who are willing to stop taking calcium supplements, if any and to restrict consumption of high calcium food to 600mg (two dairy servings) per day
* subjects with a high probability of compliance with study procedures and test article consumption
* subjects willing and able to follow protocol guidelines and schedules and complete diaries
* subjects who are likely to abstain from taking unathorized supplements or participating in any other clinical trial or experimental treatment during this trial
* subjects with normal gastrointestinal digestion and absorption

Exclusion Criteria:

* subjects who have a history of inflammatory arthritis, gout, pseudogout, Paget's disease, seizure disorder, insulin dependent diabetes mellitus, uncontrolled hypertension, unstable cardiovascular disease, active hepatic or renal disease, active cancer and/or HIV infection
* subjects who are non-ambulatory or bedridden due to osteoarthritis
* subjects who are dependent on prescription drugs to control pain
* subjects on any other clinical trial or experimental treatment in the past 3 months
* subjects who are pregnant, lactating or at risk of becoming pregnant
* subjects who have received : intramuscular corticosteroid injection or systemic corticosteroid administration within 4 weeks prior to study enrollment, intra-articular corticosteroid injection within 2 months prior to study enrollment or intra-articular hyaluronic acid injection within 4 months prior to study enrollment.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2006-01; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
WOMAC scores (pain, stiffness, mobility, total score)
6 minute walking distances
Active and Passive range of motion (goniometer measurements)
NSAID usage
Rescue medication (acetaminophen) usage

SECONDARY OUTCOMES:
DXA scans for bone mineral density
CRP levels
Lipid profiles
the safety/toxicology measurements including a chemistry profile (including serum calcium)
complete blood counts
adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Minnesota Applied Research Center, Edina, Minnesota, United States

REFERENCES:
- [Background] Frestedt JL, Walsh M, Kuskowski MA, Zenk JL. A natural mineral supplement provides relief from knee osteoarthritis symptoms: a randomized controlled pilot trial. Nutr J. 2008 Feb 17;7:9. doi: 10.1186/1475-2891-7-9. PMID 18279523
- [Derived] Frestedt JL, Kuskowski MA, Zenk JL. A natural seaweed derived mineral supplement (Aquamin F) for knee osteoarthritis: a randomised, placebo controlled pilot study. Nutr J. 2009 Feb 2;8:7. doi: 10.1186/1475-2891-8-7. PMID 19187557